CLINICAL TRIAL: NCT06292195
Title: Effects of Vitamin D on Health Promotion During Pregnancy and Its Impact on Prematurity-Related Outcome Indicators in the Alentejo Region
Brief Title: Effects of Vitamin D on Health Promotion During Pregnancy and Its Impact on Prematurity-Related Outcome
Acronym: VitDTracking
Status: Recruiting | Type: Observational
Sponsor: University of Évora (Other)
Collaborators: Comprehensive Health Research Center (Other); Unidade Local De Saúde Do Norte Alentejano (Other); Unidade local de Saúde do Baixo Alentejano (Unknown); Unidade Local de Saúde do Alentejo Central (Unknown); Universidade Nova de Lisboa (Other); Instituto de Engenharia de Sistemas e Computadores - Inovação e Desenvolvimento de Lisboa (INESC-ID) (Unknown)
Responsible Party: Principal Investigator, Maria Olívia Pereira Barbosa, Principal Investigator; MSc; PhD student, University of Évora
Other Study IDs: VitDTracking
Record Dates: First submitted 2024-02-19; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Vitamin D Deficiency; Pregnancy
Keywords: Vitamin D; Pregnancy; Prematurity; Genetic polymorphisms
MeSH Terms: conditions — Vitamin D Deficiency; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort VitDTracking: Group 1- Pregnant women with vitamin D Sufficiency (≥30 ng/mL)
  Interventions: Other: Exposure
- Cohort VitDTracking: Group 2 - Pregnant women with vitamin D Insufficiency (20-29 ng/mL)
  Interventions: Other: Exposure
- Cohort VitDTracking: Group 3 - Pregnant women with vitamin D Deficiency (<20 ng/mL)
  Interventions: Other: Exposure

INTERVENTIONS:
Other: Exposure — Maternal vitamin D levels during pregnancy (serum 25-hydroxyvitamin D levels)

SUMMARY:
The VitDTracking study focuses on the relevance of maternal vitamin D levels and their association with prematurity, aiming to improve maternal and child health outcomes, particularly by reducing avoidable preterm births. In Portugal, vitamin D levels during pregnancy have never been studied. Epidemiological data from other countries reveal a high prevalence of vitamin D deficiency/insufficiency, especially in pregnant women.

The hypovitaminoses prevalence remains high even with a supplementation dosage of 400 to 600 IU/day during pregnancy (dosage used in Portugal), which is considered as a suboptimal dose. This phenomenon is associated with adverse maternal and child outcomes, such as intrauterine growth restriction, preeclampsia, cholestasis, hypertension, and gestational diabetes as major causes of prematurity.

Additionally, the Portuguese population has a higher prevalence of genome alterations that confer a lower capacity to produce vitamin D from sunlight exposure. These genetic characteristics are present in about 19% of the population, representing a prevalence four times higher than the European average (19% versus 4.75%), leading to a higher predisposition to vitamin D deficiency.

DETAILED DESCRIPTION:
This observational study involves the implementation of multicenter recruitment centers. Data collection will take place in healthcare organizations in the Alentejo region (Évora, Beja, Portalegre, and Elvas) with a minimum total sample of 1000 pregnant women, integrating both primary and specialized healthcare, with local healthcare professionals, doctors, and nurses as collaborators.

The study will measure vitamin D levels during pregnancy and their impact on outcome indicators related to prematurity. The aim is to assess the impact of the prevalence of vitamin D deficiency on prematurity outcomes. This involves monitoring vitamin D levels in prenatal and postnatal surveillance, adding this biomarker to routine blood collections. Biometric and biochemical data collection will occur at two distinct time points. The first collection will take place during the first prenatal surveillance appointment, preferably in the first trimester. The second collection will occur postpartum, during the hospitalization period.

The study will also assess maternal vitamin D deficiency and associated factors in the Alentejo region. It aims to identify the existence of genetic polymorphisms related to vitamin D and assess associations with adverse clinical outcomes related to prematurity. This involves requesting genetic analysis by the local medical collaborator and collecting saliva from the pregnant woman (non-invasive method) for the study of polymorphisms in seven genes, integrating the analysis of 18 genetic variants that play a role in the metabolism, transport, degradation and downstream pathways of vitamin D. Saliva samples from pregnant women will be collected during hospitalization before or after birth.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women's living in the Alentejo region aged 16 years or older, who after disclosure and clarification of doubts, agree to participate in the study with signed informed consent.

Exclusion Criteria:

* Language barrier (lack of basic understanding of Portuguese).

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women's in the Alentejo region
Study Population: Pregnant women's in the Alentejo region
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-11-03 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Differences in the rate of Prematurity with different maternal Vitamin D levels | Blood samples will be taken from pregnant women up to the 13th week of pregnancy and then at the second collection point up to 48 hours after the birth (after participant enrollment; two collection points)
  Prematurity Rate in percentage
Differences in Birth Weight with different maternal Vitamin D levels | Blood samples will be taken from pregnant women up to the 13th week of pregnancy and then at the second collection point up to 48 hours after the birth (after participant enrollment; two collection points)
  Birth Weight in grams
Differences in Apgar Scores with different maternal Vitamin D levels | Blood samples will be taken from pregnant women up to the 13th week of pregnancy and then at the second collection point up to 48 hours after the birth (after participant enrollment; two collection points)
  Apgar Scores in Scale (<7 or ≥7)
Differences in the number of admissions to the Neonatal Intensive Care Unit with different maternal Vitamin D levels | Blood samples will be taken from pregnant women up to the 13th week of pregnancy and then at the second collection point up to 48 hours after the birth (after participant enrollment; two collection points)
  Number of admissions to the Neonatal Intensive Care Unit in percentage
Differences in the Neonatal Morbidity rate with different maternal Vitamin D levels | Blood samples will be taken from pregnant women up to the 13th week of pregnancy and then at the second collection point up to 48 hours after the birth (after participant enrollment; two collection points)
  Neonatal Morbidity rate in percentage
Differences in the Neonatal Mortality rate with different maternal Vitamin D levels | Blood samples will be taken from pregnant women up to the 13th week of pregnancy and then at the second collection point up to 48 hours after the birth (after participant enrollment; two collection points)
  Neonatal Mortality rate in percentage
Differences in the number of Neonatal Infections with different maternal Vitamin D levels | Blood samples will be taken from pregnant women up to the 13th week of pregnancy and then at the second collection point up to 48 hours after the birth (after participant enrollment; two collection points)
  Number of Neonatal Infections in percentage
Differences in the Number of Congenital Malformation diagnoses with different maternal vitamin D levels | Blood samples will be taken from pregnant women up to the 13th week of pregnancy and then at the second collection point up to 48 hours after the birth (after participant enrollment; two collection points)
  Number of Congenital Malformation diagnoses in percentage
Differences in the presence of vitamin D-related polymorphisms with different maternal levels of vitamin D | Saliva samples from pregnant women will be collected during admission to the hospital or up to 48 hours after delivery (after participant enrollment; single collection point)
  Differences will be assessed following the defined outcome indicators related to prematurity

SECONDARY OUTCOMES:
Differences in maternal vitamin D levels between the three groups/cohorts related to prematurity | Through study completion, an average of 3 months
Differences in maternal vitamin D levels between the three groups/cohorts related to birth weight | Through study completion, an average of 3 months
Differences in maternal vitamin D levels between the three groups/cohorts related to Apgar scores | Through study completion, an average of 3 months
Differences in maternal vitamin D levels between the three groups/cohorts related to admission to the Neonatal Intensive Care Unit | Through study completion, an average of 3 months
Differences in maternal vitamin D levels between the three groups/cohorts related to neonatal morbidity | Through study completion, an average of 3 months
Differences in maternal vitamin D levels between the three groups/cohorts related to neonatal mortality | Through study completion, an average of 3 months
Differences in maternal vitamin D levels between the three groups/cohorts related to neonatal infections. | Through study completion, an average of 3 months
Differences in maternal vitamin D levels between the three groups/cohorts related to the diagnosis of congenital malformations | Through study completion, an average of 3 months
Differences in the presence of vitamin D-related polymorphisms between the three groups/cohorts associated with prematurity | Through study completion, an average of 3 months
Differences in the presence of vitamin D-related polymorphisms between the three groups/cohorts associated with birth weight | Through study completion, an average of 3 months
Differences in the presence of vitamin D-related polymorphisms between the three groups/cohorts associated with Apgar scores | Through study completion, an average of 3 months
Differences in the presence of vitamin D-related polymorphisms between the three groups/cohorts associated with admission to the Neonatal Intensive Care Unit. | Through study completion, an average of 3 months
Differences in the presence of vitamin D-related polymorphisms between the three groups/cohorts associated with neonatal morbidity | Through study completion, an average of 3 months
Differences in the presence of vitamin D-related polymorphisms between the three groups/cohorts associated with neonatal mortality | Through study completion, an average of 3 months
Differences in the presence of vitamin D-related polymorphisms between the three groups/cohorts associated with neonatal infections | Through study completion, an average of 3 months
Differences in the presence of vitamin D-related polymorphisms between the three groups/cohorts associated with the diagnosis of congenital malformations | Through study completion, an average of 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Maria OP Barbosa, MSc; PhD student, Principal Investigator — University of Évora; Dulce Cruz, PhD, Principal Investigator — University of Évora; André Rosário, PhD, Principal Investigator — Universidade Nova de Lisboa; Marta Silvestre, PhD, Principal Investigator — Universidade Nova de Lisboa; Ana T Freitas, PhD, Principal Investigator — Instituto de Engenharia de Sistemas e Computadores - Inovação e Desenvolvimento de Lisboa (INESC-ID)
Locations (3):
- Portugal (3):
  - Unidade Local de Saúde do Baixo Alentejo, Beja
  - Unidade Local de Saúde do Alentejo Central - Hospital Espirito Santo de Évora, Evora
  - Unidade Local de Saúde do Norte Alentejano, Portalegre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barbosa O, Freitas AT, Silvestre MP, Moreira-Rosario A, Aguiar P, Regua AI, Madaleno T, Almeida M, Cruz D. Effects of Maternal Vitamin D Levels on Prematurity: Feasibility Study in a Multicenter Observational Pilot. Nutrients. 2025 Mar 27;17(7):1160. doi: 10.3390/nu17071160. PMID 40218918